CLINICAL TRIAL: NCT02022449
Title: Stress Management Intervention for At-Risk Mothers of Children With Cancer
Brief Title: Stress Management Intervention for Mothers of Children With Cancer
Acronym: CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO10040081
Record Dates: First submitted 2013-11-27; First posted 2013-12-27 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Stress; Depression
Keywords: Maternal depression; Maternal psychosocial stress and distress; Maternal health outcomes; Social support; Pediatric cancer
MeSH Terms: conditions — Depression; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): participants only complete assessments
- Stress management (Experimental): Cognitive Behavioral Stress management Coping enhancement strategies Progressive muscle relaxation Guided imagery relaxation skills Deep breathing relaxation skills Social support
  Interventions: Behavioral: Stress management

INTERVENTIONS:
Behavioral: Stress management — Cognitive behavioral stress management Cognitive and emotionally focused coping enhancement strategies Progressive muscle relaxation Social support Strategies for parenting a child with cancer
  Arms: Stress management

SUMMARY:
To explore maternal biological (activation of the hypothalamic-pituitary-adrenal axis) and behavioral (smoking, sleep behavior, exercise and alcohol use) pathways of intervention-related decreases in inflammation. Hypothesis: The intervention group will show decreased levels of cortisol and improved health behaviors from pre- to post-intervention when compared with the control group. We will also explore whether intervention-related changes in these parameters predict symptoms of illness. Exploratory Aim 2. To explore psychological pathways of intervention-related decreases in distress among mothers, including the perception of social support and the use of behavioral coping strategies that are components of the intervention. Hypothesis: Increases in perceived social support and use of active behavioral coping strategies will be associated with intervention-related decreases in symptoms of depression, anxiety and psychological stress.

ELIGIBILITY:
Inclusion Criteria:

* biologic, adoptive, or legal guardian mothers of children (birth to 17 years) who are within 6 weeks of being newly diagnosed with any cancer, with the exception of a central nervous system (CNS) cancer or early stage lymphoma, recruited from the Division of Hematology and Oncology, Children's Hospital of Pittsburgh (CHP)
* no reported clinical history of psychotic or bipolar illness, neurological disorder (stroke, transient ischemic attacks, Parkinson's disease, multiple sclerosis) or chronic disease known to influence immune function, including cardiovascular disease, cancer [within the past 2 years], or autoimmune disease
* not taking medications that might alter responses to questionnaires or indices of immune function (including major sedatives or glucocorticoid, anti-inflammatory, anti-retroviral, or immunosuppressant medication)
* fluency in English (i.e., have commonly used English in everyday speaking and reading for at least 10 years)
* is at least 18 years of age
* not working nightshifts exclusively.

Exclusion Criteria:

* mothers of children with CNS cancers due to our belief that a psychosocial intervention tailored more specifically to the unique stressors inherent in this diagnosis is warranted
* mothers of children with early stage lymphomas will be excluded because of their child's brief/mild treatment course
* mothers whose child is older than 17 years will not be eligible; the upper age limit (17 years) was established based on referral patterns at the CHP hematology/oncology department.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
change in Maternal depression is being assessed, the Beck Depression Inventory ( BDI), the Perceived Stress Scale (PSS) and other measures assessing maternal depression will be used | baseline, 2 weeks post intervention, 6 months post intervention
  maternal depression

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Ewing, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Marsland AL, Long KA, Howe C, Thompson AL, Tersak J, Ewing LJ. A pilot trial of a stress management intervention for primary caregivers of children newly diagnosed with cancer: preliminary evidence that perceived social support moderates the psychosocial benefit of intervention. J Pediatr Psychol. 2013 May;38(4):449-61. doi: 10.1093/jpepsy/jss173. Epub 2013 Jan 21. PMID 23341547
- [Derived] Lindsay EK, Inagaki TK, Walsh CP, Messay B, Ewing LJ, Marsland AL. Stress-Related Inflammation and Social Withdrawal in Mothers of a Child With Cancer: A 1-Year Follow-Up Study. Psychosom Med. 2022 Feb-Mar 01;84(2):141-150. doi: 10.1097/PSY.0000000000001037. PMID 34935760
- [Derived] Marsland AL, Walsh CP, Cleary JL, Vaisleib AD, Farrell C, Woods WC, Tersak JM, Wright A, Ewing LJ. Efficacy of a Stress Management Intervention for Mothers of Children with Cancer. J Pediatr Psychol. 2020 Jul 24:jsaa058. doi: 10.1093/jpepsy/jsaa058. Online ahead of print. PMID 32705121